CLINICAL TRIAL: NCT01157273
Title: Psychophysiological and Vocal Affections in Subjects Submitted to a Public Speaking Mock Test
Brief Title: Evaluation of Physiological and Vocal Parameters in Volunteers of Both Genders Submitted to an Anxiogenic Task
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Associação Fundo de Incentivo a Psicofarmacologia (Unknown)
Responsible Party: Anna Alice Figueiredo de Almeida, Universidade Federal da Paraiba
Other Study IDs: CEP/UNIFESP 0707/05; 142932/2006-0 (Other: CNPq)
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Anxiety; Communication
Keywords: Behavior; Anxiety; Communication; Voice
MeSH Terms: conditions — Anxiety Disorders; Communication; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High Anxiety (HA) group: 13 participants of both genders, 19-42 years old, with no history of psychiatric disorders and scores above 41 in STAI-Trait
- Low Anxiety (LA) group: 11 participants of both genders, 19-42 years old, with no history of psychiatric disorders and scores below 41 in STAI-Trait

SUMMARY:
Objective: To assess whether the anxiety caused by a task considered anxiogenic, Simulated Public Speaking (SPS) test, would change the responses of healthy individuals regarding physiological and vocal parameters. Method: The sample comprised 30 participants of both genders, 19-42 years old, with no history of psychiatric disorders. The score in the STAI-Trait enabled investigators to assign participants to two groups: LOW ANXIETY (LA) and HIGH ANXIETY (HA). The investigators evaluated physiological parameters (heart rate, skin conductance, temperature in the extremities, electromyogram of the frontal muscle and salivary cortisol) and vocal parameters (vocal self-evaluation, quality of life in voice and vocal symptoms and signs) BEFORE, DURING and AFTER the SPS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years
* Volunteers with no psychiatric history and diagnosis of vocal problem
* Have a minimum of the average school

Exclusion Criteria:

* Chronic smokers
* Subjects with paralysis or neurological diseases
* Compromised upper airway at the time of the experiment
* User stimulants, psychotropic drugs, herbal medicines, tranquilizers, antidepressants
* Have drunk coffee or alcohol on the day of the experiment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty individuals participated in the study, being 18 (60.0%) female and 12 (40.0%) male. They were between 19 and 42 years old and their schooling ranged from fundamental school (primary and middle school) to post-graduation.
  All the volunteers were in good health, had no history of psychiatric problems or alcohol and/or drug abuse, and did not report any vocal problems. Subjects excluded from the sample were chronic smokers; had paralysis or neurological diseases; had problems in the upper airways or allergic rhinitis at the moment of the experiment; used stimulant, psychotropic, anxiolytic, phytotherapic or antidepressant substances, and those who had ingested alcohol or coffee on the day of the experiment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-02; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Almeida, PhD, Principal Investigator — Universidade Federal da Paraíba
Locations (1):
- José Roberto Leite, São Paulo, São Paulo, Brazil